CLINICAL TRIAL: NCT00966446
Title: Epidemiology and Prevention of MRSA Transmission in the Community
Brief Title: Epidemiology and Prevention of Methicillin Resistant Staphylococcus Aureus (MRSA) Transmission in the Community
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Pennsylvania Department of Health (Other Government); Children's Hospital of Philadelphia (Other); Milton S. Hershey Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 809899
Record Dates: First submitted 2009-08-25; First posted 2009-08-27 (Estimated); Results first posted 2016-06-29 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: MRSA - Methicillin Resistant Staphylococcus Aureus Infection
Keywords: MRSA; household; infection; colonization
MeSH Terms: conditions — Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Unsupervised Decolonization (Experimental): Households undergo decolonization for MRSA. The intervention includes applying Mupirocin ointment twice daily for the first 7 days of study enrollment as well as using Hibliclens body wash twice total (on day 1 and day 7 of study enrollment) according to the instructions provided.
  Interventions: Drug: Unsupervised Decolonization
- Supervised Decolonization (Experimental): Households undergo decolonization for MRSA. The intervention includes applying Mupirocin ointment twice daily for the first 7 days of study enrollment as well as using Hibliclens body wash twice total (on day 1 and day 7 of study enrollment) according to the instructions provided. Study staff is in contact with household members during this intervention to ensure compliance.
  Interventions: Drug: Supervised Decolonization
- No Intervention (No Intervention): Households do not undergo active MRSA decolonization protocol

INTERVENTIONS:
Drug: Unsupervised Decolonization — Households will undergo decolonization for MRSA with Mupirocin nasal ointment and Hibiclens body wash. This means that the intervention includes applying Mupirocin ointment twice daily in each nostril for the first 7 days of study enrollment as well as using Hibliclens body wash twice total (on day 1 and day 7 of study enrollment) according to the instructions provided. Households are given detailed, written instructions and are asked to fill out logs tracking compliance for each household member.
  Other Names: Experimental: Unsupervised Decolonization
  Arms: Unsupervised Decolonization
Drug: Supervised Decolonization — Households will undergo decolonization for MRSA with Mupirocin nasal ointment and Hibiclens body wash. This means that the intervention includes applying Mupirocin ointment twice daily in each nostril for the first 7 days of study enrollment as well as using Hibliclens body wash twice total (on day 1 and day 7 of study enrollment) according to the instructions provided. Households are given detailed, written instructions and are asked to fill out logs tracking compliance for each household member. In addition, households are contacted by study stuff via phone or text messages to ensure compliance, to provide reminders to household members to perform the decolonization protocol as well as to answer any question/concerns household members may have.
  Other Names: Experimental: Supervised Decolonization
  Arms: Supervised Decolonization

SUMMARY:
The overall goal of this project is to elucidate the epidemiology of MRSA transmission in the community and test an intervention to prevent MRSA transmission in this setting.

DETAILED DESCRIPTION:
The overall goals of this project are to:

1. to investigate the determinants of and evaluate potential interventions to reduce the spread of methicillin resistant Staphylococcus aureus (MRSA) infections in community settings in order to reduce the burden of this illness in the State of Pennsylvania. This objective has the following specific aims:

   * to identify host, microbiological and environmental risk factors for prolonged MRSA colonization, MRSA transmission and clinical MRSA infection among patients with MRSA skin and soft tissue infections (SSTIs) and their household contacts and to use stochastic agent-based modeling methods to quantify secondary spread of CO-MRSA in households.
   * to evaluate the impact of a decolonization intervention on MRSA infections in the household.
   * to identify immunological mechanisms underlying the ability of Streptococcus pneumoniae colonization to inhibit MRSA colonization, transmission and infection in order to identify potential future immunological targets for interventions.
2. to foster multi-disciplinary and cross-institutional collaborations and develop the infrastructure for a Center of Excellence focused on antimicrobial drug resistance research, with the capacity for activities linking basic science, epidemiological and clinical intervention studies
3. to enhance opportunities for basic and clinical research training for undergraduate and graduate students, particularly from underrepresented minorities, in order to increase the pipeline of future biomedical scientists and clinical investigators

ELIGIBILITY:
Inclusion Criteria:

* All members of a household in which the index case is treated for a skin or soft tissue infection due to MRSA. All household members must agree to participate in order for the household to be enrolled

Exclusion Criteria:

* Prior MRSA within past 6 months in the index case; age less than 6 months.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2009-09; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ebbing Lautenbach, MD, Principal Investigator — University of Pennsylvania
Locations (4):
- United States (4):
  - Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shahbazian JH, Hahn PD, Ludwig S, Ferguson J, Baron P, Christ A, Spicer K, Tolomeo P, Torrie AM, Bilker WB, Cluzet VC, Hu B, Julian K, Nachamkin I, Rankin SC, Morris DO, Lautenbach E, Davis MF. Multidrug and Mupirocin Resistance in Environmental Methicillin-Resistant Staphylococcus aureus (MRSA) Isolates from Homes of People Diagnosed with Community-Onset MRSA Infection. Appl Environ Microbiol. 2017 Oct 31;83(22):e01369-17. doi: 10.1128/AEM.01369-17. Print 2017 Nov 15. PMID 28939607
- [Derived] Cluzet VC, Gerber JS, Metlay JP, Nachamkin I, Zaoutis TE, Davis MF, Julian KG, Linkin DR, Coffin SE, Margolis DJ, Hollander JE, Bilker WB, Han X, Mistry RD, Gavin LJ, Tolomeo P, Wise JA, Wheeler MK, Hu B, Fishman NO, Royer D, Lautenbach E; CDC Prevention Epicenters Program. The Effect of Total Household Decolonization on Clearance of Colonization With Methicillin-Resistant Staphylococcus aureus. Infect Control Hosp Epidemiol. 2016 Oct;37(10):1226-33. doi: 10.1017/ice.2016.138. Epub 2016 Jul 28. PMID 27465112

RESULTS

PARTICIPANT FLOW:
Groups:
- Supervised Decolonization: Households undergo decolonization for MRSA. Intervention includes applying Mupirocin ointment twice daily for the first 7 days of study enrollment AND using Hibliclens body wash twice total (day 1 and day 7 of study enrollment) according to the instructions provided. To ensure compliance, study staff is in contact with household members.
  Supervised Decolonization: Households will undergo decolonization for MRSA with Mupirocin nasal ointment and Hibiclens body wash. Intervention includes applying Mupirocin ointment twice daily in each nostril for the first 7 days of study enrollment AND using Hibliclens body wash twice total (day 1 and day 7 of study enrollment) according to the instructions provided. Households are asked to fill out logs tracking compliance for each household member. Study staff contacts households daily (phone/text) to ensure complicane, to provide reminders to household members to perform the decolonization protocol, and to answer study question/concerns.
Period: Overall Study
Arm/Group | Unsupervised Decolonization | Supervised Decolonization | No Intervention
Started | 76 | 74 | 73
Completed | 48 | 49 | 52
Not Completed | 28 | 25 | 21

BASELINE CHARACTERISTICS:
Groups:
- Unsupervised Decolonization: This group was randomized to the following decolonization protocol: 1) 2% mupirocin ointment applied inside both nares twice daily for seven days 2) a 4% chlorhexidine gluconate (Hibiclens, Mo¨lnlycke Health Care, Norcross, Georgia) body wash, including entire skin surface, excluding face and hair, with particular attention to axillae, inguinal region, and perirectal areas, performed on both the first and the last day of mupirocin use. Subjects were asked to record performance of each step of the decolonization protocol in a journal, which was returned at the end of the period of medication use, along with any unused portion of the mupirocin and chlorhexidine gluconate body wash containers. The subjects randomized to unsupervised decolonization were instructed on the decolonization protocol during the initial interview, along with the educational instruction as described in the "no intervention" group.
- Supervised Decolonization: This group was also randomized to the decolonization protocol. In addition those randomized to supervised decolonization received daily phone calls or text messages during the decolonization protocol period in order to remind enrolled subjects to perform the indicated procedure in addition to the instruction and education received during the initial interview.
- No Intervention: Households do not undergo active MRSA decolonization protocol. The received education only. The content of the education focused on personal hygiene (hand hygiene and bathing), interrupting transmission (avoidance of shared towels, razors, etc.), and household hygiene (regular washing of linens and towels, disposal of potentially infective materials such as bandages).
- Total: Total of all reporting groups
Arm/Group | Unsupervised Decolonization | Supervised Decolonization | No Intervention | Total
Number analyzed (Participants) | 76 | 74 | 73 | 223
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 35 | 37 | 38 | 110
  Between 18 and 65 years | 39 | 35 | 32 | 106
  >=65 years | 2 | 2 | 3 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 43 | 45 | 128
  Male | 36 | 31 | 28 | 95
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 5 | 4 | 15
  Not Hispanic or Latino | 68 | 67 | 68 | 203
  Unknown or Not Reported | 2 | 2 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 41 | 47 | 47 | 135
  White | 32 | 20 | 20 | 72
  More than one race | 1 | 1 | 1 | 3
  Unknown or Not Reported | 2 | 5 | 4 | 11
Region of Enrollment [Number; unit: participants]
  United States | 76 | 74 | 73 | 223

OUTCOME MEASURES:

1. Primary Outcome: Recurrent Infection
Description: Confirmed new MRSA infections
Time Frame: Within 6 months
Population: These study participants who self-reported re-infections of MRSA
Measure: Number; unit: participants
Groups:
- Unsupervised Decolonization: Mupirocin topical to nares twice daily x7 days; Chlorhexidine bath on Days 1 and 7
- Supervised Decolonization: Mupirocin topical to nares twice daily x7 days; Chlorhexidine bath on Days 1 and 7 with daily call/text message reminders
- No Intervention: No decolonization agents
Arm/Group | Unsupervised Decolonization | Supervised Decolonization | No Intervention
Number analyzed (Participants) | 48 | 49 | 52
participants | 1 | 3 | 1

2. Primary Outcome: First Two Consecutive Sampling Periods Completed
Description: Subjects who returned samples for at least the first two consecutive sampling periods were included in analysis
Time Frame: Within 2 months
Population: These subjects sent in two consecutive swab samples starting with their first follow-up time point.
Measure: Number; unit: participants
Arm/Group | Unsupervised Decolonization | Supervised Decolonization | No Intervention
Number analyzed (Participants) | 48 | 49 | 52
participants | 48 | 49 | 52

3. Secondary Outcome: Time to Clearance of Methicillin-resistant Staphylococcus Aureus (MRSA) Colonization
Description: Surveillance cultures negative for two consecutive sampling periods; date of clearance determined as midpoint between date of last positive surveillance culture and first negative surveillance culture.
Time Frame: Within 6 months
Population: Subjects who returned samples for at least the first two consecutive sampling periods were included in analysis, as this was necessary to determine clearance of MRSA colonization
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Unsupervised Decolonization | Supervised Decolonization | No Intervention
Number analyzed (Participants) | 48 | 49 | 52
days | 23 [17 to 29] | 23 [17 to 29] | 19 [15 to 33]

ADVERSE EVENTS:
Time Frame: 1 week
Description: Serious adverse events include:
  * Death
  * Life threatening adverse experience
  * Inpatient hospitalization/prolongation of existing hospitalization
  * Persistent disability/incapacity
  * Medical event (may not be life threatening/require immediate hospitalization) but may require medical/surgical intervention to prevent a serious adverse event.
Arm/Group | Unsupervised Decolonization | Supervised Decolonization | No Intervention
Serious Adverse Events (participants affected / at risk) | 5/76 | 7/74 | 4/73
Other Adverse Events (participants affected / at risk) | 17/76 | 29/74 | 0/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Unsupervised Decolonization (N=76) | Supervised Decolonization (N=74) | No Intervention (N=73)
heart disease (Cardiac disorders) | 0 (0) | 1 (1) | 3 (3) — This adverse event was both unrelated and unanticipated; participants had multiple chronic conditions including: CHF, PE, infarction, Afib, DM with neuropathy, HTN, CKD, Cutaneous lymphoma; inpatient hospice.
Anorexia nervosa (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
homocide (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
inflammatory bowel (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
cancer (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
hypertension (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
cancer (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
hemmorage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
abscess (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Unsupervised Decolonization (N=76) | Supervised Decolonization (N=74) | No Intervention (N=73)
runny nose (General disorders) | 4 (4) | 3 (3) | 0 (0) — subject reported a drippy nose
abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
burning (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0) — burning feeling on the skin
Broken bone (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — broken ankle
feel sick (General disorders) | 1 (1) | 4 (4) | 0 (0) — subject reported feeling ill
nasal congestion (General disorders) | 0 (0) | 6 (6) | 0 (0)
headache (General disorders) | 1 (1) | 0 (0) | 0 (0)
sore throat (General disorders) | 0 (0) | 2 (2) | 0 (0)
common cold (General disorders) | 1 (1) | 0 (0) | 0 (0)
fever (Infections and infestations) | 5 (5) | 1 (1) | 0 (0)
flu (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
itching (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0)
irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0)
sneezing (General disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes